CLINICAL TRIAL: NCT01541631
Title: Epidemiology of Human Immunodeficiency Virus (HIV-1) and Schistosoma Mansoni Co-infections and Its Impact on Anthelminthic Treatment Outcome Among HIV-1 Infected Individuals in Fishing Communities in Mwanza Region, Northwestern Tanzania.
Brief Title: A Study of Co-infections of HIV-1 and Schistosoma Mansoni and Its Impact on Praziquantel Treatment Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of Health and Allied Sciences (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); University of Cambridge (Other)
Responsible Party: Principal Investigator, Humphrey Mazigo, Msc, MPH, Epidemiology of Human Immunodeficiency Virus (HIV-1) and Schistosoma mansoni co-infections and its impact on anthelminthic treatment outcome among HIV-1 infected individuals in fishing communities in Mwanza region, Northwestern Tanzania., Makerere University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 087540; 00005856/2011 (Other: Makerere University College of Health Sciences)
Record Dates: First submitted 2012-02-20; First posted 2012-03-01 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Anemia; Intestinal Helminthiasis; Intestinal Schistosomiasis; Human Immunodeficiency Virus I Infection; Hematologic Diseases; Opportunistic Infections
Keywords: Human Immunodeficiency Virus-1; Schistosoma mansoni; Anemia; Immune response; Opportunistic infections; Tanzania
MeSH Terms: conditions — Anemia; Intestinal helminthiasis; Schistosomiasis mansoni; Hematologic Diseases; Opportunistic Infections; Schistosomiasis | interventions — Praziquantel; Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HIV-1 co-infected with schistosoma mansoni (Experimental): HIV-1 patients co-infected with Schistosoma mansoni
  Interventions: Drug: Praziquantel and Albendazole
- HIV-1 positive individuals with negative S. mansoni (No Intervention): HIV-1 positive individuals with negative Schistosoma mansoni
  Interventions: Drug: Praziquantel and Albendazole
- Schistosoma mansoni positive but HIV-1 negative (Experimental): Schistosoma mansoni positive individuals but HIV-1 negative to be compared with HIV-1 co-infected with Schistosoma mansoni individuals
  Interventions: Drug: Praziquantel and Albendazole
- HIV-1 and Schistosoma mansoni negative (No Intervention): Individuals with no HIV-1 and S. mansoni infections
  Interventions: Drug: Praziquantel and Albendazole

INTERVENTIONS:
Drug: Praziquantel and Albendazole — Praziquantel Tablet - 40mg/kgBWT given once Albendazole Tablet - 400mg once
  Other Names: DISTOCIDE; ZENTEL
  Arms: HIV-1 co-infected with schistosoma mansoni
Drug: Praziquantel and Albendazole — Praziquantel- 40mg/kgBWT Albendazole - 400mg once
  Other Names: DISTOCIDE; ZENTEL
Drug: Praziquantel and Albendazole — Praziquantel- 40MG/KG ONCE Albendazole - 400mg once
  Other Names: DISTOCIDE; ZENTEL
  Arms: HIV-1 co-infected with schistosoma mansoni; HIV-1 positive individuals with negative S. mansoni; Schistosoma mansoni positive but HIV-1 negative

SUMMARY:
In this study, it is hypothesized that helminth infections modulate immune responses against HIV-1 infection resulting into increased HIV-1 multiplication, faster progression to AIDS and increased episodes of AIDS-related opportunistic infections. Furthermore, the effect of helminth infections on progression of HIV-1 infection is dependent on helminth infection intensity, host background immunity, nutritional status, demographic factors and socio-economic status. Also, treatment of helminth infections using praziquantel and albendazole among HIV-1 infected individuals will lead to reduction in HIV-1 viral loads, improvement of CD4+ counts, CD4+/CD8+ ratio and Hb levels, improved weight gain and reduction of episodes of HIV-1 related opportunistic infections. In addition, HIV-1 infection is associated with poor anthelminthic treatment outcome as compared to non-HIV infected individuals

DETAILED DESCRIPTION:
The proposed study has the main objective to investigate the epidemiology of HIV-1 and Schistosoma mansoni co-infections and assess their association and progress of HIV positive individuals co-infected with S. mansoni. The study will also assess the impact of praziquantel treatment on S. mansoni related morbidities in co-infected HIV positive individuals with S. mansoni in Fishing villages, northwest Tanzania. The study is designed as a community based intervention trial, which consist of cross-sectional survey at the initial baseline survey followed by intervention trials. The initial baseline survey will include 2000 participants from the two villages. The objective of the survey is to determine the prevalence of HIV-1 infection and haemoglobin levels. Also, the socio-economic, demographic characteristics, individual behaviour in relation to HIV-1 and helminth transmission are recorded. In addition, the location and altitude of each household will determined using a hand-held Garmin GPSmap 60CSX, which has an accuracy of ± 5m. After initial survey, study participant will be grouped into 2 groups, one HIV-1 infected group and HIV-1 uninfected group. Blood sample for examination of CD4+, CD4+/CD8+ and HIV-1 viral loads will be obtained from HIV-1 positive participants every month for a period of six month. After 6 month of prospective longitudinal survey, the first follow-up survey of the recruited study participants will be conducted with the objective of determining prevalence and intensity of human intestinal schistosomiasis and other helminth infections. Other infections will also be examined, includes malaria and viral hepatitis. Furthermore, S. mansoni induced morbidity will be examined using ultrasonography. A blood sample will also be obtained for all HIV-1 positive patients, from which CD4+, CD4+/CD8+ and HIV-1 viral loads will be examined. In the same survey, individuals who tested HIV-1 negative at baseline will also be screened for HIV. After the first follow-up survey, three groups will be formed, Group A- individuals co-infected with HIV-1 and S. mansoni (N=270); Group B- individuals infected with HIV-1 but S. mansoni negative (N=180) and Group C- HIV-1 negative but S. mansoni positive (N=1320) (Figure 2). All individuals who will be infected with S. mansoni and other helminth detected in the study irrespective of HIV-1 serostatus will be treated with praziquantel (40mg/kg) and albendazole (400mg). At six to eight weeks after mass treatment, a second survey will be conducted in the recruited participants aiming at determining cure rates of S. mansoni after chemotherapy with praziquantel. The third survey will be conducted 12 month after the first follow-up survey with the aim of determining the change in CD4+, CD4+/CD8+, HIV-1 viral loads, HIV-1 progression and reversibility of the S. mansoni related liver morbidity after praziquantel

ELIGIBILITY:
Inclusion Criteria:

* Permanent residents and those who have lived in the village for more than 2 years.
* HIV-1 positive individuals only those with CD4+ ≥ 400 cells/μl

Exclusion Criteria:

* HIV-1 positive individuals with CD4+ < 350 cells/μl,
* Those who are on antiretroviral therapy (ARV)
* Pregnant women are excluded.
* Participants with chronic diseases such as leukemia, tuberculosis and viral hepatitis

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2000 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
The impact of Praziquantel in HIV-1 individuals co-infected with Schistosoma mansoni | 12 month follow-up
  * Impact of praziquantel treatment on CD4+,CD4+/CD8+, HIV-1 viral loads haemoglobin level, reversibility of liver pathology and occurance of opportunistic infection
  * Prevalence of co-infections of HIV-1 and Schistosoma mansoni
  * Prospective longitudinal association between HIV-1 and S. mansoni, and the progression of HIV to AIDS, according to S. mansoni infection status.

SECONDARY OUTCOMES:
Efficacy of praziquantel | 12 months
  * Cure rates
  * Reductions of infections intensities

CONTACTS AND LOCATIONS:
Overall Officials: Humphrey D Mazigo, Principal Investigator — Makerere University
Locations (2):
- Tanzania (2):
  - Ilemela District, Mwanza, Lake Victoria Zone
  - National Institute for Medical Research, Mwanza, Mwanza, Lake Victoria Zone